CLINICAL TRIAL: NCT01405859
Title: Neuroimaging to Elucidate the Mechanism of Tic Resolution in Tourette Syndrome
Brief Title: MRI Study of Tic Remission in Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Shprecher, Assistant Professor, Neurology, University of Utah
Other Study IDs: 39432
Record Dates: First submitted 2011-05-27; First posted 2011-07-29 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Tourette Syndrome
Keywords: Tourette; tic; Tourette's; Tourette syndrome; Tourette's syndrome
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TS controls: 10
- Non TS Controls: 11
- TS remission: 0

SUMMARY:
Doctors provide a ray of hope to children and their parents with the knowledge that, for most patients, symptoms of Tourette syndrome improve by the time they are young adults. The investigators do not know why some improve and others do not. This study is designed to help answer that question. The investigators will use magnetic resonance imaging (MRI) techniques to test whether individuals who experience improvement of their Tourette's (tic remission) have more mature brain connections than those who do not.

DETAILED DESCRIPTION:
One of the most interesting aspects of Tourette syndrome is a virtual remission of tics by early adulthood in about half of patients. Information is needed to clarify the mechanism of tic remission in order to guide development of better treatments for this disabling condition. For this cross-sectional study, 10 individuals with tic remission and 10 individuals with persistent Tourette syndrome are being recruited for a one-time study visit. 10 neurologically normal (non-TS) controls have also been recruited to obtain control neuroimaging data. All participants will complete a study questionnaire and a 60-minute MRI procedure. Sequences used to compare the groups will be volumetric, diffusion tensor, resting state functional connectivity MRI and MR spectroscopy. Our primary hypothesis is that the pattern of functional connectivity in individuals with tic remission will be more mature than that of those with persistent tics. Secondary hypotheses tested will explore whether the other modalities can be used to differentiate tic remission from persistent TS.

ELIGIBILITY:
Inclusion Criteria:

All subjects: males aged 18-35 with history of Tourette syndrome and at least moderately disabling tics during childhood.

Persistent Tourette's subjects: history of disabling tics during childhood but no longer taking tic suppressing drugs.

Tic remission subjects: no longer experiencing any disability (even social discomfort) from tics. Must have had sustained improvement of tics for at least 3 years.

Normal controls: no longer recruiting.

Exclusion Criteria:

Tourette's subjects still taking tic suppressing drugs are excluded. Also excluded are any patients with a condition (such as a pacemaker, recent tattoo, implantable metal device, or claustrophobia) that could make the MRI examination unsafe.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adult males (aged 18-35) with a history of Tourette syndrome, including at least moderate disability from tics during childhood.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Resting state functional connectivity | Participants come in for a one-time visit. All participants will be enrolled by July 2012. Data will be analyzed by Sept 2012.
  Quantitative measurements of integrated voxel-by-voxel blood oxygen level dependent fMRI time-series data will be compared between activated regions. Cross-correlation coefficients will be computed following band-pass filtering of data for evaluation of frequency-dependent contributions to correlation using standard functional connectivity techniques. Similar correlation analysis will be performed with signal from pulse oximetry and respiratory effort to evaluate for confounding stimulus-correlated physiological noise.

SECONDARY OUTCOMES:
Magnetic resonance spectroscopy | Participants come in for a one-time visit. All participants will be enrolled by July 2012. Data will be analyzed by Sept 2012.
  For each subject a central voxel within the anterior cingulate will be used as the region of interest. Peaks for substances of interest will be compared between each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: David Shprecher, Principal Investigator — Neurology
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3983677/ — Final Study Results, Published in Tremor and Other Hyperkinetic Disorders